CLINICAL TRIAL: NCT01799655
Title: Does Vitamin D Deficiency Associated With Hypercoagulability & Increased Thrombin Generation?
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: Vitamin D deficiency
Record Dates: First submitted 2013-02-06; First posted 2013-02-27 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2013-02

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cardiovascular disease is the most common cause of mortality and morbidity worldwide. Recently, a growing body of evidence has identified Vitamin D deficiency as a potential risk factor for cardiovascular disease. Therefore, there is an increasing interest to explore the mechanism in which vitamin D deficiency affect the cardiovascular system.

The investigators want to examine the relationship between serum vitamin D levels and the coagulation status in the subjects. The applied the calibrated automated thrombogram (CAT) to assess thrombin generation in plasma as a measure of overall thrombotic activity, and thus to suggest a mechanism that may explain the link between vitamin D deficiency and cardiovascular disease.

Our study population are going to include 100 patients from the internal departments in Emek hospital, who present with chest pain but without acute coronary syndrome (ACS). The investigators will take blood samples from the subjects to measure the serum vitamin D levels and the generation of thrombin. The patients will be divided into four groups according to the level of vitamin D to evaluate the effect of vitamin D levels in the blood on coagulability and thrombotic activity in these patients.

ELIGIBILITY:
Inclusion Criteria:

•hospitalized patient with diagnosed of chest pain

Exclusion Criteria:

•recent Myocardial ischemia - (in the last 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patient
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
thrombin generation levels and endogenous thrombin potentials | 4 month
  measuring the thrombin generation and endogenous thrombin potential by the calibrated automated thrombogram (CAT)

CONTACTS AND LOCATIONS:
Overall Officials: Mazen elias, prof, Principal Investigator — haemek medical center
Locations (1):
- Haemek medical center, Afula, Israel